CLINICAL TRIAL: NCT04855812
Title: The Efficacy of Upper Extremity Wearable Robotic Orthosis on Improving Upper Extremity Motor Function and Activities of Daily Living in Persons With Spinal Cord Injury
Acronym: MyoMo in SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: D-1028-18
Record Dates: First submitted 2020-02-03; First posted 2021-04-22 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: SCI - Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- MyoPro (Experimental): Receiving MyoMo training in-clinic and at home for 6-weeks
  Interventions: Device: MyoMo
- Myo-SB (Active Comparator): Receiving MyoMo training in-clinic and using their prescribed static brace (or others) at home for 6-weeks
  Interventions: Other: Myo-SB
- Control (Active Comparator): Receiving conventional therapy/training in-clinic and using their prescribed static brace (or others) at home for 6-weeks
  Interventions: Other: Control

INTERVENTIONS:
Device: MyoMo — To evaluate the usefulness of an upper extremity (UE) assistive device, called (MyoPro) in improving upper extremity activities in people with incomplete spinal cord injury (iSCI).
  Arms: MyoPro
Other: Myo-SB — To evaluate the usefulness of an upper extremity (UE) assistive device, called (MyoPro) in improving upper extremity activities in people with incomplete spinal cord injury (iSCI).
  Arms: Myo-SB
Other: Control — To evaluate the usefulness of an upper extremity (UE) assistive device, called (MyoPro) in improving upper extremity activities in people with incomplete spinal cord injury (iSCI).
  Arms: Control

SUMMARY:
To evaluate the usefulness of an upper extremity (UE) assistive device, called (MyoPro) in improving upper extremity activities in people with incomplete spinal cord injury (iSCI)

DETAILED DESCRIPTION:
The study will take me approximately 10 weeks from the time of consent. This includes initial screening visit, a baseline assessment, and a follow-up visit (after 6 weeks of therapy). The baseline and follow up visit will include 2 separate testing sessions, each session will last approximately 2 hours. I will also participate in approximately 3 training sessions per week for 6 weeks. Each training session will last approximately 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Be between ages 18-80.
* Be able to activate biceps & triceps brachii, and forearm muscles with sufficient muscle signal amplitude as determined by the physical/ occupational therapist.
* Be diagnosed with SCI (iSCI (ASIA Impairment Scale (AIS) C and D, (C1-C8)) and be at least 1-year post injury.
* Be medically stable.
* Be able to follow directions for the tasks of the study and to communicate in English with the study staff.
* Continue to take all prescribed medication (e.g. oral or via pump baclofen) without any dosing changes.
* Be able to tolerate functional tasks for 60min with intermittent rests without excessive fatigue.
* Have some visible muscle contraction (with or without range of motion) on their upper extremity as determined by study staff.
* Have full passive range of motion for elbow flexion and extension as determined by study staff.

Exclusion Criteria:

* Have excessive pain in the upper extremity that limits my receiving rehabilitation therapy.
* Have excessive spasticity: Patients with modified ashworth scale (MAS) of 2 and higher at the wrist or 3 at the elbow joints as determined by study staff.
* Be participating in any experimental rehabilitation or drug studies.
* Have history of neurologic disorder other than SCI.
* Have other conditions or circumstances that, in the opinion of the investigators, would preclude safe and/or effective participation, including severe sensory deficits, skin conditions, and/or other conditions that may be contradicted for myoelectric Myo-Pro use.
* Have difficulty following multiple step directions.
* Have severe problems with thinking and understanding or psychiatric problems that might limit my ability to do training.
* Have skin issues that would prevent wearing the Myo-Pro device.
* Have had history of recurrent epilepsy, seizure or convulsion
* Have a past or current history of treated ringing in the ears known as tinnitus or severe hearing problems.
* Study staff and physician will review my medications to determine if I am taking any drugs that would increase my risk of having a seizure while undergoing brain stimulation. If I am taking such a medication I will not be enrolled in this study.
* Because of potential risk to the fetus, women of child bearing potential will be required to have a pregnancy test before they can enroll in this study. If I am female, and have a positive pregnancy test, I will not be enrolled.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-27 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Range of motion of hands and arms | Approximately 10 weeks
  Movement of upper extremity is measured using small sensors that are able to record joints' angles. These sensors are placed on participant's skin via double sticky tape.
  Participants will be asked to move their hand and forearm while the elbow, wrist and hand joint angles are measured.
Muscle strength measurement | Approximately 10 weeks
  during movements of upper extremities muscle strength is measured using small and light weight surface electromyography sensors which are placed on the participant's skin via double stick tape.
  Participants will be asked to move their hand and forearm while the muscle strength is measured.
Brain signals measurement | Approximately 10 weeks
  Measurements of brain signals is done using a cap and electrodes that would be placed on the participant's head using surface electrodes.
  Participants will be asked to move their extremities while brain signals are measured.
GRASSP | Approximately 10 weeks
  Assessment of the Hand in Tetraplegia Using the Graded Redefined Assessment of Strength Sensibility and Prehension Upper Extremity Function in Persons with Tetraplegia Relationships Between Strength, Capacity and the Spinal Cord Independence Measure.
  Total score's minimum and maximum values are between 0 to 116 and higher scores indicate better/improved outcomes.
Spasticity measurement | Approximately 10 weeks
  Spasticity measurements of upper and lower extremities using the Modified Ashworth scale (MAS).
  The MAS scores range between 0 to 4. A higher score signifies larger level of spasticity and a lower score indicates smaller level of spasticity. scores are as follows:
  0: No increase in muscle tone
  1. Slight increase in muscle tone 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of motion
  2. More marked increase in muscle tone through most of the range of motion.
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
CUE-Q | Approximately 10 weeks
  The Capabilities of Upper Extremity Test (a list of questionnaire based evaluation).
  Scores range between 0 to 4, and higher scores indicates better ability outcome for reaching or lifting the upper limb.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided